CLINICAL TRIAL: NCT03286296
Title: A First-in-Human, Multicenter, Open-label, Phase 1 Dose-Escalation Study of LZM009 in Subjects With Advanced Solid Tumors
Brief Title: LZM009 to Treat Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LZM009-001
Record Dates: First submitted 2017-09-08; First posted 2017-09-18 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LZM009 (Experimental)
  Interventions: Biological: LZM009,recombinant humanized anti-PD-1 monoclonal antibody for injection

INTERVENTIONS:
Biological: LZM009,recombinant humanized anti-PD-1 monoclonal antibody for injection — LZM009 doses of 1, 3, and 10 mg/kg will be administrated intravenously on day 1 and 29 and every 3 weeks thereafter until disease progression or intolerable toxicity, withdrawal of consent, or end of study

SUMMARY:
To assess the safety and tolerability of IV administered LZM009 in subjects with advanced solid tumors who have progressed or are non-responsive to available therapies.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Histologically or cytologically confirmed solid malignancy.
2. Male or non-pregnant, non-lactating female patients age ≥18 years.
3. Locally advanced or metastatic disease that is refractory to standard therapy [note for patients with NSCLC patients with activating ALK translocation or EGFR mutations must have been treated and failed appropriate therapy], or for which there is no standard available therapy.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
5. Subject with a life expectancy of ≥ 12 weeks.
6. Adequate hematologic function as indicated by

   1. Platelet count ≥ 100,000/mm3
   2. Hemoglobin ≥ 9.0g/dL
   3. Absolute neutrophil count (ANC) ≥1000/uL Note: Use of growth-factors to maintain ANC criterion (within 28 days prior to the first dose of study drug and within 28 days after day 1 of Cycle 1) is not permitted.
7. Adequate renal and liver function as indicated by:

   1. Serum creatinine ≤ 1.5 x upper limit of normal (ULN); if serum creatinine is >1.5 x ULN, creatinine clearance must be ≥ 50 mL/min either by calculation or by measured 24-hour urine collection
   2. Total bilirubin ≤1.5 x ULN; If Gilbert's Syndrome may have Bilirubin> 1.5 x ULN
   3. Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤3 x ULN of institution's normal range; for patients with known liver metastases, AST and ALT may be ≤ 5 x ULN.
   4. Coagulation: aPTT and PT≤ 1.3 x ULN
8. Patients with brain metastases are eligible if clinically controlled that is defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function & no evidence of CNS disease progression as determined by CT or MRI within 21 days prior to the first dose of study drug.
9. Willingness to use contraception by a method that is deemed effective by the investigator by both males and female patients of child bearing potential (postmenopausal women must have been amenorrheal for at least 12 months to be considered of non-childbearing potential) and their partners throughout the treatment period and for at least three months following the last dose of study drug.
10. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the patient prior to any study-specific procedures).
11. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

To be eligible for entry into the study, the subject must not meet any of the exclusion criteria listed below:

1. Receiving concurrent anti-cancer therapy or investigational therapy (chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, targeted therapy, biologic therapy, (with the exception of hormones for hypothyroidism, estrogen replacement therapy, or LHRH agonists required to suppress serum testosterone levels).
2. Patients who have experienced a Grade 3 or higher toxicity related to prior PD-1/PD-L1 treatment.
3. Prior anticancer therapy less than 21 days of study entry, or 5 half-lives, whichever is shorter.
4. Steroid therapy for anti-neoplastic intent within 7 days prior to the first dose of study drug.
5. Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to ≤ Grade 1.
6. Known bleeding diathesis/disorder unless controlled.
7. Recent history of non-chemotherapy induced thrombocytopenia associated bleeding within 1 year prior to first dose of study drug.
8. Have active immune thrombocytopenic purpura (ITP), active autoimmune hemolytic anemia (AHA), or a history of being refractory to platelet transfusions (within 1 year prior to the first dose of study drug).
9. Serious gastrointestinal bleeding within 3 months.
10. Received a biologic (G-CSF, GM-CSF or erythropoietin) within 28 days prior to the first dose of study drug and within 28 days after the first dose.
11. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days before the planned first dose of study drug. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease. Ophthalmologic, nasal and intra-articular injections or steroids are acceptable.
12. Failure to recover adequately, as judged by the investigator, from prior surgical procedures. Patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry.
13. Unstable angina, myocardial infarction, or a coronary revascularization procedure within 180 days of study entry.
14. Neurologic instability per clinical evaluation due to tumor involvement of the central nervous system (CNS). Patients with CNS tumors that have been treated, are asymptomatic and who have discontinued steroids (for the treatment of CNS tumors) for>28 days may be enrolled.
15. Positive laboratory test for HBsAg or anti-HCV. Patients with anti-hepatitis B core antibody are eligible if negative for HBsAg; patients positive for anti-HCV may be enrolled if negative by nucleic acid amplification test.
16. Has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening.
17. Any diagnosis of autoimmune disease. Subjects with hypothyroidism stable on hormone replacement, adrenal insufficiency on steroid replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment are permitted to enroll.
18. Grade 3 or higher pneumonitis or neuropathy during previous treatment with immunotherapy.
19. Diagnosis of fever and neutropenia within 1 week prior to study drug administration.
20. Uncontrolled concurrent illness including, but not limited to: serious uncontrolled diabetes (blood glucose > 250 mg/dL), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
21. Patient has received a live, attenuated vaccine within 28 days of planned start of study therapy.
22. Known allergies, hypersensitivity, or intolerance to protein-based therapies or with a history of any significant drug allergy (e.g., anaphylaxis, hepatotoxicity, immune-mediated thrombocytopenia or anemia), or to LZM009 recipients (refer to Investigator's Brochure).
23. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 21 days or 5 half-lives, whichever is shorter, before the start of study treatment, the exception of participants in the follow-up phase.
24. Any other condition or circumstance of that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Determine number of patients experiencing dose limiting toxicities | Day 1 through Day 28
  And frequency and severity of DLT at LZM009 doses of 1mg/kg, 3mkg/kg and 10mkg/kg at 28 days after the first dose.
Determine Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) | 17 months
  Determination of MTD and RP2D is dependent on number of cohorts and patients experiencing DLT.
Number of patients experiencing clinical or laboratory adverse events as a measure of safety and tolerability | Screening to 28 days after last treatment administration, or until drug related toxicities have resolved, whichever is later; or earlier than 28 days should the patient commence another anti-cancer therapy in the meantime, approximately 17 weeks.
  Safety variables include incidence and severity of treatment emergent adverse events (TEAEs) and immune-related AEs (irAEs), vital signs measurements, clinical laboratory values and ECGs as determined by CTCAEv4.03.

SECONDARY OUTCOMES:
Characterize the pharmacokinetics (PK) profiles of LZM009 in blood specimens of subjects with at least 1 dose | Predose, 0 h, 2 h, 6h, 24h, days 3, 8, 15 and 22 post infusion of cycle 1; predose of cycle 2 and 3; pre-dose, 0 h, 2 h, 6h, days 8, and 15 post infusion of cycle 4 and predose of every other cycle after Cycle 5(one cycle=21 days except Cycle 1=28 days).
Characterize the immunogenicity profiles of LZM009 in blood specimens of subjects with at least 1 dose | Predose on C1D1, C2D1, C4D1, and at predose of every other cycle after Cycle 5, thereafter for the first 12 months, and 28 days after the last dose(one cycle=21 days except Cycle 1=28 days).
  Presence of anti-LZM009 antibodies/neutralizing anti-LZM009 antibodies (nAbs) and effect on PK of LZM009.
Assess preliminary anti-tumor activity of LZM009 in subjects with advanced solid tumors | 17 months
  Overall response rate (ORR) by the Response Criteria in Solid Tumors (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - START Midwest, Grand Rapids, Michigan
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas